CLINICAL TRIAL: NCT06395168
Title: IMPAC: Integrated Maternal Postpartum Appointment Combination in Mayo Clinic Health System Northwest Wisconsin
Brief Title: Mayo Clinic Health System Northwest Wisconsin Integrated Maternal Postpartum Appointment Combination
Acronym: IMPAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Melissa A. Thompson, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-012862
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Lactation and Newborn visit (Active Comparator): This arm is the intervention where the newborn visit with the pediatric provider is within a lactation consultant visit for a breastfeeding newborn and mother.
  Interventions: Other: Combined Newborn and Lactation Visit
- Separate Lactation and Newborn visit (No Intervention): This is current state of care in which a newborn visit is separate and apart from a Lactation Consultation.

INTERVENTIONS:
Other: Combined Newborn and Lactation Visit — See Arm/Group Description
  Arms: Combined Lactation and Newborn visit

SUMMARY:
The purpose of this study is to explore whether combining the first post-hospital newborn provider visit and lactation consultation into a single appointment can enhance rates of successful breastfeeding initiation and continuation at predefined intervals (e.g., one week, one month, two months, three months, four months, six months, and 12 months postpartum).

DETAILED DESCRIPTION:
This interventional, comparative effectiveness study investigates the impact of integrating the first newborn outpatient provider and lactation consultant visits, potentially reducing appointments for new mothers while ensuring early lactation support. The outcomes, including breastfeeding continuation rates and maternal satisfaction, will be measured against the conventional separate visit model. The ultimate goal is to prolong breastfeeding duration, enhance care quality, improve efficiency, and enrich patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Mothers aged greater than or equal to 18 years.
* Mothers who are able to provide informed consent for participation in this study.
* Mothers registered as patients at Mayo Clinic Health System Northwest Wisconsin.
* Mothers who have given birth within the past four days prior to enrollment into this study.
* Mothers who intend to breastfeed their newborns.
* Mothers who are willing and able to participate in this study.
* Mothers who are able to communicate in English.
* Mothers with the ability to connect to the internet and complete electronic data collection.

Exclusion Criteria:

* Mothers who are unable or unwilling to provide informed consent for participation in this study.
* Mothers less than 18 years of age.
* Mothers unable to complete study procedures or follow-up visits.
* Mothers with medical complications that could interfere with breastfeeding (e.g., breast reduction).
* Mothers who have no intention to breastfeed their newborns.
* Mothers who are unwilling to follow up with lactation.
* Infants who have already had their first postpartum outpatient provider visit.
* Pre-term infants (less than 37 weeks).
* Special care admission greater than two days.
* Length of stay or anticipated LOS greater than four days.
* Transfer to an outside facility.
* Inability to communicate in English.
* When slots are no longer available.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Difference of breastfeeding rates with a combined lactation/newborn visit versus separate visits. | Duration of the study (expected 1 year)
  Looking for the difference of breastfeeding continuation between the intervention and control group. Hypothesis is higher breastfeeding rates in the combined lactation/newborn visit.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Thompson, CNP, DNP, APNP, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials